CLINICAL TRIAL: NCT06105333
Title: Fidgety Movements of Preterm Neonates Included in COSGOD III - Ancillary Retrospective Observational Study to COSGOD III Trial
Brief Title: Fidgety Movements of Preterm Neonates Included in COSGOD III
Acronym: Figdety_Ms
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Figdety Movements - COSGOD III
Record Dates: First submitted 2023-10-06; First posted 2023-10-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Preterm; General Movements; Fidgety Movements; Near Infrared Spectroscopy; Neurological Outcome
Keywords: near-infrared spectroscopy; preterm neonates; preterm birth; cerebral injury; cerebral oxygenation; resuscitation; neurological outcome; fidgety movements; general movements
MeSH Terms: conditions — Premature Birth; Brain Injuries | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIRS Group: Preterm neonates less than 32 weeks gestation were randomly assigned to standard care plus cerebral oxygen saturation monitoring with a dedicated treatment guideline (NIRS-group) during immediate transition (first 15 minutes after birth) and resuscitation.
  Interventions: Procedure: standard care plus cerebral oxygen saturation monitoring with a dedicated treatment guideline
- Standard Care Group: Preterm neonates less than 32 weeks gestation were randomly assigned to standard care (control-group) with routine monitoring during immediate transition (first 15 minutes after birth) and resuscitation.

INTERVENTIONS:
Procedure: standard care plus cerebral oxygen saturation monitoring with a dedicated treatment guideline — CrSO2 (Cerebral regional oxygen saturation) monitoring was visible to the clinical team with the same SpO2 target as in the control group. If SpO2 (oxygen saturation) remained between the 10th and 90th centiles and within local limits, and crSO2 was <10th centile according to published reference ranges, FiO2 (fraction of inspired oxygen) was increased by 10-20% every 60 seconds or respiratory support was started or increased. If crSO2 remained >10th centile for >60 seconds or if rSO2 was >90th centile,FiO2 was reduced by 10-20% or respiratory support was adjusted accordingly. If there was a history of blood loss or clinical signs of blood loss, intravenous fluids (10 mL/kg) were considered.
  Groups: NIRS Group

SUMMARY:
The evidence on the effects of clinical care with cerebral NIRS (Near-infrared spectroscopy) monitoring on short term neurological outcome, displayed by fidgety movements between six to 20 weeks post term, are still uncertain.

Two centers (Graz and Innsbruck), who participated in the COSGOD III trial, routinely performed GMA between 37+0 to 42+0 weeks of corrected age (writhing movements) and between six to 20 weeks post term (fidgety movements).

Aim of the present study is therefore to assess in neonates, who were included into the COSGOD III trial, in a retrospective observational study routinely performed fidgety movements between six to 20 weeks of corrected age after discharge.

The investigators hypothesise that the preterm neonates in the intervention group of the COSGOD III trial show better survival and short term neurological outcome, displayed by normal fidgety movements, compared to neonates in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates included in the COSGOD III trial
* Death
* Routinely performed fidgety movement (FM) analysis between six to 20 weeks post term

Exclusion Criteria:

* Neonates without FM analysis between six to 20 weeks post term

Max Age: 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates < 32 weeks of gestational age included in COSGOD III trial in Graz and Innsbruck are eligible to be included in this ancillary study.
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Short-term outcome | Between six to 20 weeks post term in surviving preterm neonates
  Combined outcome of survival with normal Fidgety movement analysis. Outcome defined as good (survival with normal fidgety movements) or poor (death, abnormal/absent of fidgety movements). Mortality is assessed by medical documentation system.
  Fidgety movement assessements were performed by video recording of sequences of at least three minutes. Fidgety movements were documented by clinical staff trained and certified for GMA. FMs were as either normal or abnormal, whereby abnormal FMs are further divided into two categories: absent or abnormal.

SECONDARY OUTCOMES:
Interventions during resuscitation | First 15 minutes after birth
  Interventions during the first 15 minutes after birth include n (%) of supplemental oxygen, respiratory support, chest compression, caffeine, adrenaline, surfactant, volume. These data were documented in the eCRF.
Interventions during the first 24 hours after birth | First 24 hours after birth
  Interventions during the first 24 hours after birth include n (%) of surfactant, no respiratory support, non-invasive ventilation and mechanical ventilation. These data were documented in the eCRF.
Neonatal morbidity at term age | Between birth and term age
  Neonatal morbidities include n (%) of IVH (any grade), cystic PVL, IRDS, culture proven sepsis, NEC, BPD, ROP and PDA with interventions. These data were documented in the eCRF.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, Prof., Principal Investigator — Division of Neonatology, Medical University of Graz, Austria
Locations (2):
- Austria (2):
  - Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck

IPD SHARING:
Plan to Share IPD: No